CLINICAL TRIAL: NCT06446011
Title: Potential Effects of Non-surgical Endodontic Treatment on Periapical Healing, Inflammatory Markers, and Kidney Function Indicators in Chronic Kidney Disease Patients With Apical Periodontitis- Interventional Study.
Brief Title: Effects of RCT on Periapical Healing, Inflammatory Markers, and Kidney Function Indicators in CKD Patients With AP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Himanshi Verma
Record Dates: First submitted 2023-12-07; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2023-11

CONDITIONS: Apical Periodontitis; Chronic Kidney Diseases
MeSH Terms: conditions — Periapical Periodontitis; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic kidney disease group (Experimental): Root canal treatment will be performed in teeth with apical periodontitis in chronic kidney disease patients and change in PAI score, eGFR and systemic markers will be checked.
  Interventions: Procedure: root canal treatment in Ckd patients
- Healthy group (Active Comparator): Root canal treatment will be performed in teeth with apical periodontitis in healthy patients and change in PAI score and systemic markers will be checked
  Interventions: Procedure: root canal treatment in healthy patients

INTERVENTIONS:
Procedure: root canal treatment in Ckd patients — root canal treatment in teeth with apical periodontitis to observe periapical healing , and change in eGFR ,blood urea and creatinine and HSCRP
  Arms: Chronic kidney disease group
Procedure: root canal treatment in healthy patients — root canal treatment in teeth with apical periodontitis to observe periapical healing and change in HSCRP
  Arms: Healthy group

SUMMARY:
The purpose of this prospective study is to determine the effect of non-surgical root canal treatment in chronic kidney disease patients and healthy patients with apical periodontitis.

DETAILED DESCRIPTION:
It has been found that there is an association between prevalence of odontogenic infection and systemic diseases. An elevated level of systemic cytokines has been observed in conjunction with both AP and CKD . The proinflammatory status and impaired immune response associated with systemic diseases (chronic kidney disease ) can affect the reparative response of the dental pulp and periapical healing. One study observed significant positive relation between number of diagnosed AP and urea serum level . A 4.35-mg/dL increase in the urea serum level could be expected per 1-unit increase in the number of teeth with AP. Improving oral health care through nonsurgical endodontic treatment(NSET) may improve the systemic inflammatory status and improve renal function.

The aim of this prospective study is to determine the effect of non-surgical root canal treatment in chronic kidney disease patients and healthy patients with apical periodontitis

1. Clinical and radiographic success rate will be considered as primary outcome, will be checked at baseline,6months,12months follow up.Periapical status will be checked according to periapical index given by Orstavik
2. Reduction in inflammatory(hsCRP) and kidney makers(serum urea , creatinine , eGFR) will be considered as secondary outcome, will be checked at baseline,3months,6months follow up.

ELIGIBILITY:
Inclusion Criteria:

1- Known patient of Chronic Kidney Disease [CKD Stages 1,2,3,4,5 with mature permanent teeth.

2. Age18year or older . 3. ≥ to 12 natural teeth (excluding 3rd molars) 4 The periapical index (PAI) was used to evaluate the periapical status patients with PAI ≥3 are included in the study.

Exclusion Criteria:

1. Patients having systemic disorders other than chronic kidney disease (e.g HIV; Diabetes mellitus; Coronary heart disease; no history of secondary hyperparathyroidism)
2. Patients with periodontitis , pocket depth and CAL>5mm( stage 3 ,4) will be excluded.
3. Pregnancy; lactation & contraceptives.
4. Patients taking antibiotics, statins, corticosteroids and aspirin which can affect the level of inflammatory markers in past one month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender matched healthy control participants to the same gender chronic kidney disease individuals will be analyzed.
Enrollment: 74 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Periapical Index(PAI) | 12MONTHS
  Periodical status will be assessed in periodical radiograph and scoring of periapical index will be done according to size and periphery of peri-apical radiolucency with coding 1 to 5

SECONDARY OUTCOMES:
eGFR | 3-6MONTHS
  BY BLOOD SAMPLE measured in mL/min/1.73m2
serum creatinine | 3-6MONTHS
  BY BLOOD SAMPLE measured in mg/dL
hs-CRP | 3-6MONTHS
  HIGH SENSITIVE C-reactive protein measured by ELISA kit in mg/L
Blood urea | 3-6MONTHS
  measured by collecting blood sample in mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: HIMANSHI VERMA, MDS, Principal Investigator — PGIDS,ROHTAK
Locations (1):
- PGIDS, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No